CLINICAL TRIAL: NCT02666703
Title: Immunomodulatory Effect of Extracorporeal Cytokine Adsorption in Cardiac Surgery
Brief Title: Extracorporeal Cytokine Adsorption in Cardiac Surgery
Acronym: IMEECCACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Gordana Taleska, MD, MSc, Spec., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARRS-RPROJ-2014-191
Record Dates: First submitted 2016-01-17; First posted 2016-01-28 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiopulmonary Bypass
Keywords: cardiac surgery; systemic inflammatory response; immunoadsorption
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study (CytoSorb) (Experimental): In the study group (20 patients) the CytoSorb filter will be installed in the CPB in a parallel circuit. An additional roller pump will drive the blood through the filter with a constant flow of 400 ml/min (max flow).
  Interventions: Device: CytoSorb
- Control (No Intervention): In the control group (20 patients) no filter will be installed on the CPB.
- Corticosteroid (Active Comparator): In the corticosteroid group (20 patients), 1 gram of methylprednisolone will be added in the priming solution of CPB machine. No filter will be installed on the CPB.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Device: CytoSorb — CytoSorb is a first-in-class extracorporeal cytokine adsorber, now approved in the European Union, and broadly indicated for use in any clinical situation where cytokines are elevated.
  Arms: Study (CytoSorb)
Drug: Methylprednisolone
  Arms: Corticosteroid

SUMMARY:
The modern era of cardiac surgery began in early 1950s with the introduction of cardiopulmonary bypass (CPB). Although it has been clearly shown that CPB is almost unavoidable for most open heart operations, an undesirable systemic inflammatory response syndrome (SIRS) is associated with its use. This complex chain of events has strong similarities with sepsis and may contribute to the development of postoperative complications and multiple organ failure (MOF). It has been shown that an excessive compensatory anti-inflammatory response (CARS) after SIRS can lead to immune paralysis and increased rate of hospital acquired infection. The balance of pro-inflammatory and anti-inflammatory mediators determines the inflammatory response and the clinical outcome. Accordingly, great efforts have been focused on therapeutic interventions aimed at reducing the inflammatory reactions during CPB, including pharmacologic strategies and modification of surgical techniques or mechanical devices. Such therapies may provide improvements in patient outcome after open heart operations. Among pharmacologic strategies is the prophylaxis with corticosteroids, which have been used during open heart surgery for more than 30 years. Many studies, both experimental and clinical, failed to produce evidence in favor of steroid treatment. As far as medical devices are concerned, the use of extracorporeal cytokine filter CytoSorb looks promising in cardiac surgery. It was recently approved by European Medicines Agency as an active treatment to fight cytokine storm.

Serum paraoxonase 1 (PON1) is a lipo-lactonase, being associated with HDL that has an anti-inflammatory role and protects against atherosclerosis. Low levels of PON1 are associated with venous graft occlusion in patients with coronary artery bypass grafting. PON1 reduces monocyte chemotaxis and adhesion to endothelial cells, leading to inhibition of the differentiation of monocytes into macrophages. The effects of cytokine adsorption therapy on PON1 are unknown.

The aim of the study is to explore the effects of extracorporeal immunoadsorption during CPB on pro-inflammatory and anti-inflammatory protective mediators and cellular immune status in cardiac surgery.

DETAILED DESCRIPTION:
Patients undergoing complex cardiac surgery with CPB (eg: combined valve and coronary bypass grafting surgery, concomitant valve surgery, surgery of the ascending aorta and aortic arch, as well as re-operations of the same type) will be enrolled in the study after giving the signed informed consent. They will be randomized into 3 groups: 1. study (CytoSorb) group, 2. control group, and 3. corticosteroid group. Immune response [TNF-alfa (tumor necrosis factor-alpha), IL(interleukin)-1, IL-6, IL-8, IL-10, complement C5a, lymphocyte cellular markers (CD64, CD163), miRNA (micro RNA), PON1 activity, as well as lipid status, hs-CRP (high sensitivity C-reactive protein), PCT (procalcitonin) and acute phase proteins, will be determined before CPB, during CPB, immediately after, 24h, 48h and 5 days after CPB. We will document demographic characteristics of patients, their preoperative medical status, as well as intraoperative data (type and duration of surgery, duration of CPB, period of ischemia, hemodynamic parameters, usage of inotropic/vasoactive therapy, insulin, fluids, blood and blood components); duration of mechanical ventilation in intensive care unit (ICU), duration of ICU stay, 30-day mortality and morbidity, as well as postoperative complications (bleeding, hemodynamic instability, impaired respiratory function, infection, worsening of renal, liver and cognitive function).

ELIGIBILITY:
Inclusion Criteria:

* Elective complex cardiac surgery (combined valve and coronary bypass grafting surgery, concomitant valve surgery, surgery of the ascending aorta and aortic arch, as well as re-operations of the same type)
* Age > 18 years

Exclusion Criteria:

* Disagreement to participate in the study
* Age < 18 years
* Pregnancy
* Emergency procedure
* Heart transplantation
* Implantation of LVAD (left ventricular assist device), RVAD (right ventricular assist device) or TAH (total artificial heart)
* Treatment with chemotherapy, immunosuppressive therapy
* Treatment with anti-leukocyte drugs or TNF-alfa blockers
* Immunocompromised patients (AIDS), leucopenia (< 4,0x109 / L)
* Clinical and/or laboratory signs of infection (CRP >2 mg/dl)
* Serum creatinine >2 mg/dl
* Bilirubin >2 mg/dl
* History of stroke
* Malnourished patients, BMI < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Evolution of pro-inflammatory and anti-inflammatory cytokines [TNF-alfa, IL-1, IL-6, IL-8 and IL-10 | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Evolution of complement C5a | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Evolution of CD 64 and CD 163 markers | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Evolution of miRNA | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Evolution of PON1, HDL and LDL | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb

SECONDARY OUTCOMES:
Changes in serum hs-CRP | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Changes in serum PCT | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Changes in white blood count | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb
Changes in serum albumin and fibrinogen | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day); only for Study group-1 h after start of CPB: 7)from blood entering CytoSorb and 8)from blood leaving CytoSorb

OTHER OUTCOMES:
Duration of postoperative mechanical ventilation | duration of ICU stay, an expected average of 2 days
Length of ICU stay | duration of ICU stay, an expected average of 2 days
Use of inotropic/vasoactive drugs and insulin | 1) before induction of anesthesia; 2)at the end of CPB; 3) at the end of surgical procedure; 4) 24 h; 5) 48 h; 6) 5th postoperative day
  assessed by the dose - mcg/kg/min for inotropic/vasoactive drugs and IU/h for insulin
Length of hospital stay | through study completion, an average of 1 year
30 days mortality | at day 30

CONTACTS AND LOCATIONS:
Overall Officials: Maja Sostaric, MD, PhD, Study Director — University Medical Centre Ljubljana; Matej Podbregar, MD, PhD, Study Director — University Medical Centre Ljubljana; Gordana Taleska, MD, MSc, Principal Investigator — University Medical Centre Ljubljana; Tomislav Klokocovnik, MD, PhD, Study Director — University Medical Centre Ljubljana
Locations (1):
- University Medical Center, Ljubljana, Slovenia

REFERENCES:
- [Derived] Taleska Stupica G, Sostaric M, Bozhinovska M, Rupert L, Bosnic Z, Jerin A, Ihan A, Klokocovnik T, Podbregar M. Extracorporeal Hemadsorption versus Glucocorticoids during Cardiopulmonary Bypass: A Prospective, Randomized, Controlled Trial. Cardiovasc Ther. 2020 Mar 27;2020:7834173. doi: 10.1155/2020/7834173. eCollection 2020. PMID 32292492